CLINICAL TRIAL: NCT05053477
Title: Ultrasound-Guided Pulsed Radiofrequency Versus Perineural Platelet Rich Plasma Injection for Treatment of Idiopathic Carpal Tunnel Syndrome, A Prospective Randomized Controlled Study
Brief Title: Radiofrequency, Perineural Injection, Idiopathic Carpal Tunnel Syndrome
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Alexandria University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 1216-4-009
Record Dates: First submitted 2021-09-11; First posted 2021-09-22 (Actual); Last update posted 2021-09-29 (Actual); Status verified 2021-01

CONDITIONS: Carpal Tunnel Syndrome
Keywords: CTS, Platelet Rich Plasma, Pulsed Radiofrequency
MeSH Terms: conditions — Carpal Tunnel Syndrome | interventions — Pulsed Radiofrequency Treatment

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Control Group (Active Comparator): Patients will receive median nerve perineural injection of bupivacaine with mehylprednisolone under ultrasound guidance
  Interventions: Drug: mehylprednisolone injection
- PRF Group (Active Comparator): Patients will receive median nerve pulsed radiofrequency (PRF) and median nerve perineural injection of bupivacaine under ultrasound guidance
  Interventions: Device: pulsed radiofrequency (PRF)
- PRP Group (Active Comparator): Patients will receive median nerve perineural injection of platelet-rich plasma (PRP) under ultrasound guidance
  Interventions: Biological: platelet-rich plasma

INTERVENTIONS:
Drug: mehylprednisolone injection — (40 mg)
  Other Names: Group A
  Arms: Control Group
Device: pulsed radiofrequency (PRF) — . PRF lesion will be carried out for 120 seconds at a 2 Hz frequency and pulse width of 20 ms at 42°C
  Other Names: Group B
  Arms: PRF Group
Biological: platelet-rich plasma — 2 ml of PRP
  Other Names: Group C
  Arms: PRP Group

SUMMARY:
Aim of the study The aim of the study is to evaluate the role of pulsed radiofrequency versus platelet rich plasma injection in treatment of idiopathic mild to moderate carpal tunnel syndrome Patients will be classified into three equal groups using randomized closed envelop method into three groups.

Control Group ( n=25):Patients will receive median nerve perineural injection of bupivacaine with mehylprednisolone under ultrasound guidance.

PRF Group ( n=25):Patients will receive median nerve pulsed radiofrequency (PRF) and median nerve perineural injection of bupivacaine under ultrasound guidance PRP Group (n=25): Patients will receive median nerve perineural injection of platelet-rich plasma (PRP) under ultrasound guidance

Measurements (will be done before the procedure, one week ,two month and four months after procedure except SNCV and serum CRP and TNF α (tumor necrosis factor alpha)will be done before the procedure and after four months only):

1. VAS (visual analogue pain scale)
2. BCTQ (Boston carpal tunnel Questionnaire)
3. Degree of paresthesia tested by Reverse Phalen's test.
4. CSA (cross sectional area)0 of the median nerve will be measured by the same pain therapist involved in the study.
5. SNCV (nerve conduction velocity study): performed by same physiotherapist not involved in the study before and after intervention.
6. Serum Tumor necrosis factor alpha (TNF α).
7. C-reactive protein (CRP)
8. Complications will be recorded and managed. Items 1,2 and 3 will be measured by a pain therapist not involved in this study

DETAILED DESCRIPTION:
Introduction Carpal Tunnel Syndrome (CTS) is the most common form of entrapment neuropathy. CTS is defined as a symptomatic compression neuropathy of the median nerve at the level of the wrist, characterized physiologically by evidence of increased pressure within the carpal tunnel and decreased function of the nerve at this level.

Diagnosis of CTS is mainly a clinical one based on the history and physical examination by Tinnel's test Phanel's test and Reverse Phalen's test.The Reverse Phalen's test is more appropriate clinical test for truly compressing the carpal tunnel and provoking symptoms of CTS The gold standard of diagnosis is nerve conduction velocity study (SNCV) and ultrasonography. SNCV is highly specific and it rules out neuropathies and demyelinating disease but it has a considerable false negative rate of 10-20% . Ultrasonography has high sensitivity (89%) and specificity (83%) for the diagnosis of CTS.

Median nerve cross-sectional area (CSA) is used for the assessment and the grading of median nerve pathology. While patients hold their wrists in a neutral position with the palm up and fingers semi-extended, the CSA of the median nerve will be measured in ellipse adjusted to maximum transverse and anteroposterior diameter at the proximal inlet of the carpal tunnel at the level of the pisiform bone. The normal CSA is 9 mm2. The cross-section area cutoff points that discriminate between different grades of CTS severity are 10-15 mm2 for mild to moderate symptoms, and >15 mm2 for severe symptoms PRF treatment is well established intervention technique for treatment of CT.Although the mechanism of action of PRF is not yet known but it has been postulated that PRF has a neuromodulatory effect as it modifies the neuronal membranes and selectively targets the small diameter C and A -ᶑ fibers PRP is autologous fraction of human blood that encompasses a bigger concentration of platelets than baseline levels of blood. PRP contains platelet degradation production the form of multiple growth factors such as are transforming growth factor beta (TGF beta),vascular endothelial growth factor (VEGF) platelet-derived growth factor (PDGF), and epithelial growth factor (EGF). PRP therapies aim to enhance the self-healing ability of human body, by exposing the injured tissue to a high concentration of autologous growth factors. Increased Schwann cell proliferation, myelinization, axonal regeneration, and better nerve healing after injury have been reported.

The immune system has increasingly been implicated in numerous neurological disorders. Patients with CTS have adaptive changes in the homeostasis of memory T cells and an increase in systemic inflammatory response modulating cytokines/chemokines. Which is a prominent feature of neuroinflammation and elevated levels of certain cytokines such as TNFα, IL-6 (interlukin 6), and IL-1β, have been demonstrated in patients with painful peripheral neuropathies.

Aim of the study The aim of the study is to evaluate the role of pulsed radiofrequency versus platelet rich plasma injection in treatment of idiopathic mild to moderate carpal tunnel syndrome

Plan of the study Inclusion criteria

* Patients aged (30-50) years of both gender.
* Patients with mild to moderate idiopathic CTS.
* Patient who are failed to respond to conservative treatment (such as splint, medications, physical therapy) for at least three months.

Exclusion criteria Severe CTS and secondary CTS.

Patients will be classified into three equal groups using randomized closed envelop method into three groups.

Control Group ( n=25):Patients will receive median nerve perineural injection of bupivacaine with mehylprednisolone under ultrasound guidance.

PRF Group ( n=25):Patients will receive median nerve pulsed radiofrequency (PRF) and median nerve perineural injection of bupivacaine under ultrasound guidance PRP Group (n=25): Patients will receive median nerve perineural injection of platelet-rich plasma (PRP) under ultrasound guidance

METHODS

Assessment and Preparation:

Patients will be then assessed by:

Detailed medical and surgical history taking. Clinical examination for median nerve by Reverse Phalen's test, Tinel's tests and Boston Carpal Tunnel Syndrome Questionnaire (BCTQ) Cross-sectional area (CSA): The median nerve will be identified using a 38 mm,L25x ,13-6 MHz, linear array transducer with a portable, bedside Ultrasound unit (Sonosite S-Nerve ,Sonosite Inc.,USA). The probe will be inserted in transversve direction at proximal crease of hand.

Nerve conduction velocity study (SNCV)

Laboratory investigations via venous blood sample:

* Platelet count.
* Random blood sugar.
* Coagulation profile (PT,PTT, INR).
* C-reactive protein (CRP)
* Immune test :Serum Tumor necrosis factor alpha (TNF α). All the procedures and the tests including VAS and BCTQ questionnaire will be explained to all the patients.

All patient will be admitted to day case unit then they will be transferred to block room , On arrival to the block room, patients will be connected to the standard monitoring (Drager Infiniti Gamma Patient Monitor) to display the following:

* Three lead Electrocardiogram
* Peripheral arterial oxygen saturation
* Non-invasive arterial blood pressure All patient will receive intravenouse sedation via peripheral line as midazolam with dosage range: 0.5 to 2 mg over ≥2 minutes; will repeat every 2 to 5 minutes as needed; titrate to clinical effect; maximum total dose: 5 mg.

In patient randomized to PRP group, 10 ml of whole blood will be freshly collected from each patient on citrated tube.The tubes will be initially centrifuged using (Electric centrifuge, model 800,China ) at 3000 rpm for 3 minutes. The supernatant plasma will be collected in another sterile plain tube and will be centrifuged again at 4000rpm for 15 minutes. The supernatant platelet poor plasma (PPP) will be removed leaving 2 ml of PRP on sediment (platelet pellet) which will be suspended by gently shaking the tube.

Intervention: With the palm facing upwards and the wrist joint in slight extension, the median nerve will be identified at the inlet of the carpal tunnel at the level of the pisiform bone using linear array transducer of bedside ultrasound unit. The skin will be prepared with povidone and draped in a sterile fashion, then local anesthetic infiltration using 1ml xylocaine 2% (Debocaine vial, sigma tec pharmaceutical) will be given using a 25-gauge needle.

Control Group : A 22-gauge needle of venous cannula will be gently advanced in transverse direction under ultrasound guidance using the in-plane technique via ulnar side of wrist towards the median nerve and 1ml bupivacaine 0.25% (Sunny bupivacaine vial, sunny medical group) plus 1ml (40 mg) mehylprednisolone (Solu Medrol 500mg vial, Pfizer) in total volume 2ml will be injected in perineural plane in the carpal canal.

PRF Group : After US identification of the median nerve , a 5-cm radiofrequency curved cannula with a 10-mm active tip will be inserted under ultrasound guidance using the in-plane technique in transverse direction. Using (Neurotherm NT1000, Neurotherm Inc., USA) sensory and motor stimulation will be tested after the needle tip placement near the median nerve. Responses to sensory and motor stimulation will be checked at 50 Hz, 0.5 V and at 2 Hz, 1 V respectively. PRF lesion will be carried out for 120 seconds at a 2 Hz frequency and pulse width of 20 ms at 42°C. Then 2ml of bupivacaine 0.25% will be injected perineurally.

PRP Group : A 22-gauge needle of venous cannula will be gently advanced in transverse direction under ultrasound guidance using the in-plane technique under ultrasound guidance using the in-plane technique towards the median nerve and 2 ml of PRP will be injected perineural in the carpal canal.

Post Procedure Care For Three Groups:

* Patients will be advised to apply ice on the injection site at day of intervention and modify activity as tolerated to alleviate any post injection discomfort or pain .
* Pain medication in the form of paracetamol (500mg) only will be allowed for the next 3 months if needed. The patients will be instructed to stop analgesics 48hr before visit of follow up to allow proper symptoms assessment.
* Physical therapy, splinting, or exercise will not allowed.

Measurements (will be done before the procedure, one week ,two month and four months after procedure except SNCV and serum CRP and TNF α will be done before the procedure and after four months only):

1. VAS
2. BCTQ
3. Degree of paresthesia tested by Reverse Phalen's test.
4. CSA of the median nerve will be measured by the same pain therapist involved in the study.
5. SNCV: performed by same physiotherapist not involved in the study before and after intervention.
6. Serum Tumor necrosis factor alpha (TNF α).
7. C-reactive protein (CRP)
8. Complications will be recorded and managed. Items 1,2 and 3 will be measured by a pain therapist not involved in this study.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged (30-50) years of both gender.
* Patients with mild to moderate idiopathic CTS.
* Patient who are failed to respond to conservative treatment (such as splint, medications, physical therapy) for at least three months

Exclusion Criteria:

* Severe CTS and secondary CTS

Ages: 30 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 75 (Estimated)
Dates: Start 2018-09-01 (Actual); Primary Completion 2022-11-30 (Estimated); Study Completion 2023-12 (Estimated)

PRIMARY OUTCOMES:
Evaluate the role of pulsed radiofrequency versus platelet rich plasma injection in treatment of idiopathic mild to moderate carpal tunnel syndrome | four month
  We will evaluate the median nerve by NCV to all participant
Evaluate effect of pulsed radiofrequency versus platelet rich plasma injection on pain mediators | four month
  We will measure the level of TNF to all participant

SECONDARY OUTCOMES:
Pain relief assessment | four month
  We will evaluate pain relieve by visual analogue pain scale (0_10 where 0 is no pain and 10 is maximum pain)to all participant
Numbness relief assessment | four month
  assess the numbness by Boston Carpal Tunnel Questionnaire to all participant

CONTACTS AND LOCATIONS:
Overall Officials: engy yousry, MD, Study Director — STAFF
Locations (2):
- Egypt (2):
  - Medical Research Institute, Alexandria, Alex
  - Medical Research Institute, Alexandria

IPD SHARING:
Plan to Share IPD: Yes
we share the researches to be available for general knowledge
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: after finishing the thesis for life long
Access Criteria: Digital Library Unit-Alexandria University
URL: https://www.alexu.edu.eg/